CLINICAL TRIAL: NCT04925128
Title: Effects of Moderate Physical Activity on Diabetic Adhesive Capsulitis: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RCRS/SPT/01240
Record Dates: First submitted 2021-03-31; First posted 2021-06-14 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Adhesive Capsulitis of Shoulder
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: two groups with randomization. Assignment; treadmill walking
Who Masked: Participant
Masking Description: single participant according to study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Moderate Physical Activity + Conventional Physical Therapy) (Experimental): Conventional Physical Therapy group recieved Hot pack and TENS for 10 minutes at the affected shoulder. Passive shoulder mobilizations were performed initially at pain free range in anterior, posterior, and inferior direction (10 reps x 1 set). Shoulder rolls, pendulum stretch, cross body arm stretch and towel stretch (10 reps x 1 set) were actively performed by the patient with-in limits of pain
  Moderate physical activity on treadmill, brisk walk was performed 5 days a week for 30 minutes at 4 mph speed (3-6 METs) with warm up for a 5 minutes at low speed and then at the end speed was also decreased for a 5 minutes
  Interventions: Other: Moderate Physical Activity + Conventional Physical Therapy
- Control (Conventional Physical Therapy) (Active Comparator): Conventional Physical Therapy group recieved Hot pack and TENS for 10 minutes at the affected shoulder. Passive shoulder mobilizations were performed initially at pain free range in anterior, posterior, and inferior direction (10 reps x 1 set). Shoulder rolls, pendulum stretch, cross body arm stretch and towel stretch (10 reps x 1 set) were actively performed by the patient with-in limits of pain
  Interventions: Other: Conventional Physical Therapy

INTERVENTIONS:
Other: Moderate Physical Activity + Conventional Physical Therapy — Hot pack and TENS for 10 minutes at the affected shoulder. Passive shoulder mobilizations were performed initially at pain free range in anterior, posterior, and inferior direction (10 reps x 1 set).
  Shoulder rolls, pendulum stretch, cross body arm stretch and towel stretch (10 reps x 1 set) were actively performed by the patient with-in limits of pain Moderate physical activity on treadmill, brisk walk was performed 5 days a week for 30 minutes at 4 mph speed (3-6 METs) with warm up for a 5 minutes at low speed and then at the end speed was also decreased for a 5 minutes
  Arms: Experimental (Moderate Physical Activity + Conventional Physical Therapy)
Other: Conventional Physical Therapy — Hot pack and TENS for 10 minutes at the affected shoulder. Passive shoulder mobilizations were performed initially at pain free range in anterior, posterior, and inferior direction (10 reps x 1 set).
  Shoulder rolls, pendulum stretch, cross body arm stretch and towel stretch (10 reps x 1 set) were actively performed by the patient with-in limits of pain
  Arms: Control (Conventional Physical Therapy)

SUMMARY:
The study is designed to determine the effects of moderate physical activity on adhesive capsulitis in patients with uncontrolled diabetes mellitus.

DETAILED DESCRIPTION:
This study aims to investigate the effect of additional Physical activity programmes in patients with Diabetic Frozen Shoulder (DFS).

Physical activity can help people with diabetes achieve a variety of goals, including increased cardiorespiratory fitness, increased vigour, improved glycemic control, decreased insulin resistance, improved lipid profile, blood pressure (BP) reduction and maintenance of weight loss Frozen shoulder syndrome, also known as adhesive capsulitis, is a clinical entity that refers to a stiff and painful shoulder causing major functional impairment. It affects women more than men, and is mostly associated with diabetes mellitus as a systemic condition. . Frozen shoulder may be either primary idiopathic or secondary to a systemic disease, such as diabetes mellitus.

The adoption and maintenance of physical activity are critical for blood glucose management and overall health in individuals with diabetes. In this Position Statement, we provide a clinically oriented review and evidence based recommendations regarding physical activity and exercise in people with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria :

1. The male and female physically active with uncontrolled diabetic (>6.5% HBA1c) patients those taking medicine to controlled it from more than 3 years.
2. The age of the participants will be between 40 to 65-years,
3. having stage 1 or 2 adhesive capsulitis (AC) with a capsular pattern included in the study.

Exclusion Criteria:

1. The patients with history of shoulder dislocation
2. Lower limb injury,
3. Diabetic foot ulcer,
4. Diabetic neuropathy,
5. Acute or chronic heart disease,
6. Rheumatologic disorder
7. Mobility disorder and post-surgical or trauma related patients will be excluded during the screening.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Average Blood Glucose Level | From baseline to 6th week
  The average blood glucose level for past two to three months will be measured throgh the HbA1c test, also known as the haemoglobinA1c . The normal range for the hemoglobin A1c level is between 4% and 5.6%. Between 5.7% and 6.4%indicates pre-diabetes. 6.5% or higher indicates diabetes. Validity (r=0.96 and 0.99) and reliability (r=0.95 and 0.97)
Shoulder Pain | From baseline to 3rd week and 6th week
  Shoulder pain will be assessed with numeric pain rating scale (NPRS), a reliable (Cronbach's α=0.94) and valid tool (CI = 0.96 to 0.98) for assessing pain
Shoulder ROMs | From baseline to 3rd week and 6th week
  Shoulder abduction, external rotation and internal rotation will be assessed with goiniometer for the degree and quality of this movement. The reliability of goiniometer for shoulder ROMs is ICC=0.94 and validity ICC=0.94.
Shoulder Functionality | From baseline to 3rd week and 6th week
  Disability of Arm, Shoulder, and Hand (DASH) questionnaire will be used to assess shoulder functionality which is considered a reliable and valid tool for upper limb function. It has been used for shoulder assessment in patients with AC. Validity and Reliability of this scale is (ICC=0.95) and (ICC=0.92) respectively

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No